CLINICAL TRIAL: NCT04986384
Title: Effect of a Topical Spray on Itch Relief in Moderate-to-severe Childhood Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. HON Kam Lun Ellis (Other)
Responsible Party: Sponsor-Investigator, Prof. HON Kam Lun Ellis, Department of Paediatrics, 6/F, Lui Chee Woo Clinical Sciences Building, Prince of Wales Hospital, Shatin, Hong Kong, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BAIS2018
Record Dates: First submitted 2021-05-29; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-05

CONDITIONS: Eczema
Keywords: itch relief; childhood; eczema; topical spray; quality of life
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Active Comparator): Patients will be instructed to use the anti-pruritic spray for four weeks starting from the day which informed consent was signed in active treatment group. A follow-up visit will be on week 2 for a mid-term review.
  Interventions: Drug: Atoderm SOS spray Aerosol 200ml
- Wait-list Control Group (Active Comparator): Patients will be instructed to start the treatment after two weeks from the day which consent was signed and for a duration of two weeks in wait-list control group. A follow-up visit will be on week 2 for a mid-term review and for the dispense of treating material.
  Interventions: Drug: Atoderm SOS spray Aerosol 200ml

INTERVENTIONS:
Drug: Atoderm SOS spray Aerosol 200ml — A bottle of 200ml topical spray was used on the eczematous skin lesions for itch relief.

SUMMARY:
Pruritus is defined as an unpleasant sensation of the skin that provoke the desire to scratch or rub. Its presence is an essential diagnostic feature. According to some European studies, 91% of patients with Atopic Dermatitis report suffering from pruritus at least once daily. And 58.1% of them experience chronic pruritus, leading to great deterioration in quality of life. Various internal and external factors may trigger pruritus. Mediators secretion such as keratinocyte-derived Thymic Stromal Lymphopoietin (TSLP) and Nerve Growth Factor (NGF) could activate nerve fibres which will eventually transmit signals to the brain causing the sensation of itching.

Although being one of the major annoying symptoms faced by patients with Atopic Dermatitis, effective anti-itching treatments are not available. There is no consistent evidence that topical antihistamines can relief itch.

Recently, a new spray named Atoderm 'SOS' is developed. The skin relief technology (by ambora extract and Epigallocatechin gallate (EGCG), associated to enoxolone) claimed to inhibit the release TSLP and NGF which eventually could reduce nerve signals to the brain for itchy feelings. Therefore, our group would like to test the efficacy of this proprietary anti-itch product with our paediatric patients using a wait-list approach as a control. It is aimed to demonstrate that the using the Atoderm 'SOS' spray topically whenever necessary can reduce the unpleasant itchy Atopic Dermatitis's symptom, improve quality of life, as well as to reduce the need for topical treatment.

ELIGIBILITY:
Inclusion Criteria:

* A pruritus frequency of more than 3 days in previous week recorded by Q1 in The Patient Oriented Eczema Measure (POEM)
* History of known moderate-to-severe eczema
* Able to read Chinese
* voluntarily willing to participate into the study by written consents endorsed by patients and their legal guardians

Exclusion Criteria:

* No history of known eczema
* Concurrently participating into another clinical trial
* History of known drug allergy
* unable to read Chinese

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
SCORing Atopic Dermatitis (SCORAD) | 4 weeks
  A questionnaire to examine the difference in eczema severity between two arms
The Patient Oriented Eczema Measure (POEM) | 4 weeks
  A questionnaire to examine the difference in eczema severity between two arms
Nottingham Eczema Severity Score (NESS) | 4 weeks
  A questionnaire to examine the difference in eczema severity between two arms
The Children's Dermatology Life Quality Index (CDLQI) | 4 weeks
  A questionnaire to examine the difference in quality of life between two arms
Pediatric Allergic Disease Quality of Life Questionnaire (PADQLQ) | 4 weeks
  A questionnaire to examine the difference in quality of life between two arms

SECONDARY OUTCOMES:
Bacterial colonization | 4 weeks
  Investigating the presence of Staphylococcus aureus
dermatological parameters on skin | 4 weeks
  Measuring the level of skin hydration, transepidermal water loss, and erythema
seromarkers | 4 weeks
  Measuring the amount of Brain-derived neurotrophic factor, anti-Staphylococcal enterotoxin B antibody, Immunoglobulin E, and complete blood counts.

CONTACTS AND LOCATIONS:
Overall Officials: Kam Lun Ellis KL Hon, MD, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Paediatrics, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The IPD involved sensitive clinical information which was regarded as patients' privacy. The overall study results could be found in published journal.